CLINICAL TRIAL: NCT01258491
Title: Double-blind, Randomized, Placebo-controlled, Single-center, 2 Treatment, 3-way Crossover Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of a Single Oral Repeated Dose of 500 mg Nicotinic Acid as Tablets in Healthy Subjects
Brief Title: Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of a Single Oral Repeated Dose of 500 mg Nicotinic Acid as Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Gerd Mikus, University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: K115
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2005-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Nicotinic Acids

INTERVENTIONS:
Drug: Nicotinic Acids

SUMMARY:
The study will be a double-blind, randomized, placebo-controlled, single-center, 2 treatment,3-way crossover to investigate the pharmacodynamics, i.e. the flush-symptom of a single oral repeated dose of 500 mg nicotinic acid in healthy subjects. Subjects will be randomly allocated to a treatment sequence - AAB, ABA or BAA. The two treatments will be:

* Treatment A: 500 mg nicotinic acid
* Treatment B: Placebo

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50 and 90 kg with a body mass index between 19 and <30 kg/m2
* No clinically relevant findings in the medical history, laboratory examinations and physical examination, especially with regard to cardiovascular system, liver function test, bilirubin values and the skin
* No clinical relevant pathological findings in electrocardiogram (ECG)
* Normal blood pressure (BP, syst. 100 to 140 mmHg, diast. 60 to 90 mmHg) and pulse rate (between 50 and 90 beats/min) in sitting position
* Voluntarily signed informed consent after full explanation of the study to the participant

Exclusion Criteria:

* Treatment with any other investigational product in the last 60 days before the day of randomization into the study
* Regular use of medication in the last 60 days before the day of randomization into the study except of oral contraceptives in female participants
* Treatment in the 60 days before the day of randomization into the study with any drug known to have a well-defined potential for toxicity to a major organ, or any substance which is known to induce or inhibit hepatic drug metabolism (including general anesthetics)
* Any drug intake (including over-the-counter remedies) in the 2 weeks before the day of randomization into the study, unless the investigator considers a drug intake to be clinically irrelevant for the purpose of this study
* Any acute or chronic illness or clinically relevant findings in the pre-study examination
* Presence, history or sequelae of gastrointestinal (e.g. peptic ulcer), liver or kidney disease, or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* History of hypersensitivity to the investigational product
* History or presence of abnormalities of the vascular bed
* History or presence of a dermatologic disease or skin lesions, particular in the area chosen for flush measurement
* History of allergy or hypersensitivity to other drugs or to food constituents
* History of other allergic diseases or hypersensitivity, unless the investigator considers it to be clinically irrelevant for the purpose of this study
* Blood donation of >400 ml in the 60 days before the day of randomization into the study
* Smoking
* Positive result in urine screen for drugs of abuse or in alcohol breath test
* Known or suspected to be drug-dependent, including consumption of >30 g alcohol per day
* Pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)